CLINICAL TRIAL: NCT00210561
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy and Safety of ULTRACET® (Tramadol HCl/Acetaminophen) for the Treatment of Acute Low Back Pain
Brief Title: A Study of the Effectiveness and Safety of Tramadol HCl/Acetaminophen Compared to Placebo in Treating Acute Low Back Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was stopped shortly after initiation due to change in strategic direction of the company; no safety concerns were observed that impacted this decision.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002863
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Back Pain; Low Back Pain
Keywords: Pain; Acute Low Back Pain; Back; Lower back
MeSH Terms: conditions — Back Pain; Low Back Pain; Pain | interventions — Ultracet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: tramadol hydrochloride , acetaminophen

SUMMARY:
The purpose of this study is to explore the pain-relieving effects and safety of Tramadol HCl/acetaminophen as compared to placebo in patients experiencing acute low back pain. Tramadol HCl/acetaminophen is approved for short-term management of acute pain. The combination of tramadol HCl/acetaminophen has been shown to be effective for the treatment of acute musculoskeletal pain. Patients who experienced at least moderate acute low back pain for 2 to 10 days before study entry will be randomized to receive either tramadol HCl/acetaminophen or placebo.

DETAILED DESCRIPTION:
Tramadol HCl/acetaminophen is approved for short-term (five days or less) management of acute pain. The combination of tramadol HCl/acetaminophen has been shown to be effective for the treatment of acute musculoskeletal pain. The current study is a multicenter, randomized, double-blind, placebo-controlled, parallel group study. Patients with acute low back pain for 2 to 10 days before study entry will be enrolled. At the screening visit, patients will complete questionnaires about their level of pain and disability. Patients will be randomized (like the toss of a coin) to receive either tramadol HCl/acetaminophen or placebo. Patients will take 2 tablets of study medication every 4 to 6 hours as needed for low back pain, but not more than 8 tablets per 24-hour period. Patients will call the Interactive Voice Response (IVR) system to complete a pain assessment prior to taking the first dose of study medication. Also starting on Day 1, patients will call the IVR system every night at bedtime for the remainder of the study, to complete assessments related to the following: low back pain and pain relief in the last 24 hours, current pain, pain interference with sleep and the number of study medication tablets and doses taken that day. The objective of this study is to compare the effectiveness and safety of tramadol HCl/acetaminophen versus placebo for the treatment of acute low back pain.

2 tramadol/acetaminophen 37.5/325 milligram oral tablets or 2 placebo tablets every 4 to 6 hours as needed for low back pain, but no more than 8 tablets per day, for 5 days, or until there is no further need for pain medication

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic with acute low back pain, with or without radiating pain no lower than the knee, for 2 to 10 days
* Average acute low back pain score in the last 24 hours of >= 5 on an 11-point scale at Visit 1
* In generally good health
* If female of childbearing potential, using an acceptable method of birth control

Exclusion Criteria:

* No use of ibuprofen, acetaminophen, or aspirin within 6 hours of the first dose of study medication
* No use of any other prescription or over-the-counter medication for pain within 24 hours of the first dose of study medication
* No use of medications for epilepsy or depression in the past 3 weeks
* No use of steroids within 3 months of study entry or any other long-term treatment with steroids
* No use of of tramadol HCl, tramadol HCl/acetaminophen, or any other oral opioid or opioid combination during the course of the current episode of acute low back pain
* No use of transcutaneous electrical nerve stimulation (TENS) unit within 2 weeks of study entry
* No use of an investigational drug in past 30 days
* No use of botulinum toxin for the treatment of back pain within 3 months
* No chronic continuous back pain or acute pain on top of chronic back pain
* No acute low back pain associated with chills or fever
* No pain below the knee
* No neurological signs, such as muscle weakness
* No risk of spinal infection
* No worsening of pain when lying down
* No history of significant medical conditions
* No need for urgent evaluation of the spine by neuroimaging
* No treatment during this episode by a chiropractor, physical therapy, massage, acupuncture, or Reiki treatments
* No current litigation over back pain
* No back pain related to a motor vehicle accident or work injury
* No pain more painful than their low back pain
* No progressive or degenerative neurological disorders
* No kidney damage
* Not pregnant or breast-feeding
* No condition that might affect the way the body absorbs or processes the study drug
* No bleeding condition
* No history of suicidal ideas or suicide attempts in the past 2 years
* No history of a major psychiatric disorder in past 6 months
* No history of drug or alcohol abuse or dependence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-03; Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Pain relief on Day 2 of treatment with study medication

SECONDARY OUTCOMES:
Analgesic scores for the entire treatment period including: pain relief across all study days, Brief Pain Inventory, Roland and Morris Disability Questionnaire, Subject Global Impression of Change at final visit

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of ULTRACET® (Tramadol HCl/Acetaminophen) for the Treatment of Acute Low Back Pain — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=495&filename=CR002863_CSR.pdf